CLINICAL TRIAL: NCT01576354
Title: A Phase IIb, Double-blind, Randomized, Mono-center, Placebo-controlled Study With Crossover Design Characterizing the Effects of Prolonged-release Fampridine Treatment on Ambulatory Function in Patients With Multiple Sclerosis Using Detailed Gait Analysis Based on Kinematic and Kinetic Parameters
Brief Title: Characterization of the Effects of Prolonged-release Fampridine on Ambulatory Function in Patients With Multiple Sclerosis
Acronym: FAMPKIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAMPKIN
Record Dates: First submitted 2012-03-22; First posted 2012-04-12 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; walking function; fampridine
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Prolonged-release Fampridine (Active Comparator)
  Interventions: Drug: Prolonged-release Fampridine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prolonged-release Fampridine — 10mg tablet twice a day (every 12 hours), orally
  Other Names: 4-aminopyridine, dalfampridine, ampyra, fampyra
  Arms: Prolonged-release Fampridine
Drug: Placebo — tablet twice a day (every 12 hours), orally (matched placebo is provided as oval-shaped, white to off-white, matrix tablets. Each tablet contains the following inactive ingredients: colloidal silicon dioxide, hydroxypropyl methylcellulose, magnesium stearate, microcrystalline cellulose, polyethylene glycol, and titanium dioxide)
  Arms: Placebo

SUMMARY:
The objective of the present investigator-initiated mono-center trial to be performed at the Department of Neurology of the University Hospital Zurich is a detailed characterization of the effects of prolonged-release fampridine on walking function of 50-70 patients with MS. In a randomized, double-blind, placebo-controlled study with cross-over design, changes of essential gait elements such as stability, coordination, correct loading, posture or endurance in addition to walking speed after treatment with prolonged-release fampridine will be investigated using a comprehensive kinematic gait analysis protocol. This protocol comprises outcome parameters ranging from very specific and sensitive biomechanical measures to clinically meaningful indicators of improved ambulatory function. Kinematic, kinetic and electromyographic gait parameters will be assessed during treadmill walking (primary outcome parameters). Changes in overground walking capacity will be investigated by means of different functional walking tests (e.g. six minute walk test). Furthermore, the patient's perception of the effects of the treatment on walking function will be evaluated by a standardized questionnaire. Changes of global ambulatory activity will be assessed (Actimeter) indicating a successful translation of improved gait (sub-)functions due to prolonged-release fampridine treatment into everyday life. The study will last for a period of 18 weeks, excluding the screening period. Based on the mechanism of action, the investigators hypothesize that treatment with prolonged-release fampridine will not only improve walking speed, but also clinically more meaningful features of walking function in patients with MS.

* Trial with medicinal product

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Male or female subjects must be 18 to 65 years old, inclusive, at the time of informed consent.
3. Must have a diagnosis of either primary progressive, secondary progressive, progressive remitting, or relapsing remitting MS as defined by the revised McDonald Committee criteria [Lublin et al. 1996; McDonald et al. 2001; Polman et al. 2005; Section 22.4, Appendix L] of at least 3 months duration.
4. Must be able to walk at least 50 meters (with or without a walking aid) at each individual 6minWT conducted pre-randomization.
5. Must have an impaired walking function demonstrated by a mild gait ataxia (Functional System (FS) score = 2 in the cerebellar system component of the EDSS) or a FS score of > 2 in the pyramidal system component of the EDSS based only on evaluation of the lower limbs (hip flexors, knee flexors, knee extensors, and ankle dorsiflexors)or a restricted ambulation (< 1h walking duration) at the Screening Visit.
6. Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.
7. Subjects must be able to understand the patient information sheet and comply with the requirements of the protocol.

Main Exclusion Criteria:

* Any history of seizure, epilepsy, or other convulsive disorder, with the exception of febrile seizures in childhood.
* Any prior treatment with anti-epileptic medications specifically prescribed for the treatment of epilepsy.
* Onset of MS exacerbation within the 60 days prior to the Screening Visit.
* Use of mitoxantrone, cyclophosphamide, rituximab, alemtuzumab, daclizumab, cladribine or any other immune suppressant (except FTY720) or antibody (except natalizumab) within 3 months prior to the Screening Visit, or scheduled use during study participation.
* Pulsed steroid treatment within the 60 days prior to the Screening Visit, or at any time during the screening period.
* Women who are pregnant or breast feeding,
* Clinically significant concomitant disease states such as renal failure, (e.g., moderate or severe renal impairment), hepatic dysfunction (e.g., acute or chronic hepatitis), cardiovascular or pulmonary disease, malignant disease (tumor, neoplasia) etc.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Contraindications to the class of drugs under study, e.g. known allergy to pyridine-containing substances.
* Any prior treatment with fampridine (4-aminopyridine; 4 AP) or 3,4-diaminopyridine in any formulation.
* Patients with an acute urinary tract infection at the Screening Visit as indicated by symptoms like painful urination/dysuria, urinary frequency, urinary urgency, pollakiuria, suprapubic pain, flank pain, costovertebral angle tenderness or fever >38°C in combination with a clinically significant pathological finding in the urine analysis (e.g., positive for leukocytes) at the Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Changed walking pattern on treadmill under fampridine treatment. | Assessment during double-blind fampridine and double-blind placebo treatment (each for 6 weeks, assessments in week 4 and 6). Averaged values from the 2 different testing sessions per treatment period will be compared.
  Electromyographic, kinematic and kinetic gait parameters describing stability, balance, posture, foot placement, loading, intra- and interlimb coordination and general dynamics of lower extremities will be recorded during treadmill walking.

SECONDARY OUTCOMES:
6 minute Walking Test | The test will be performed at all Visits (14) over a period of 18 weeks. Subjects will complete the task once per testing session/visit.
Timed 25-foot Walk test | The test will be performed 13 times over a period of 18 weeks. Subjects will complete the task four times per testing session/visit, two times with and two times without walking aids (in case walking aids are required).
Timed-Up-and-Go test | Subjects will complete the task two times per testing session/visit, once with and once without walking aids (in case walking aids are required). The task will be performed 4 times over a period of 18 weeks.
Berg Balance Scale | The subjects' performances are rated 4 times over a period of 18 weeks.
Dynamic Gait Index | The performance is rated 4 times over a period of 18 weeks.
LEMMT | Lower Extremity Manual Muscle Test will be performed 4 times over a period of 18 weeks.
  modified British Medical Research Council (BMRC) manual muscle test: hip flexors, knee flexors, knee extensors, and ankle dorsiflexors
Actimeter | The device will be worn for 14 days during each double-blind treatment periods (two 6-weeks-periods).
12-item MS Walking Scale | Subjects are asked to complete the standardized questionnaire 4 times over a period of 18 weeks.
Fatigue Questionnaire (WEIMuS) | Subjects are asked to complete the standardized questionnaire at each visit except the Screening Visit (i.e., 13 times) over a period of 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Linnebank, MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Zorner B, Hostettler P, Meyer C, Killeen T, Gut P, Linnebank M, Weller M, Straumann D, Filli L. Prognosis of walking function in multiple sclerosis supported by gait pattern analysis. Mult Scler Relat Disord. 2022 Jul;63:103802. doi: 10.1016/j.msard.2022.103802. Epub 2022 Apr 10. PMID 35487034
- [Derived] Weller D, Filli L, Meyer C, Lorincz L, Linnebank M, Weller M, Curt A, Zorner B. Impaired speed-dependent modulation of the gait pattern in multiple sclerosis. J Neurol. 2020 Oct;267(10):2998-3007. doi: 10.1007/s00415-020-09965-3. Epub 2020 Jun 4. PMID 32500374
- [Derived] Filli L, Werner J, Beyer G, Reuter K, Petersen JA, Weller M, Zorner B, Linnebank M. Predicting responsiveness to fampridine in gait-impaired patients with multiple sclerosis. Eur J Neurol. 2019 Feb;26(2):281-289. doi: 10.1111/ene.13805. Epub 2018 Oct 7. PMID 30171655
- [Derived] Filli L, Zorner B, Kapitza S, Reuter K, Lorincz L, Weller D, Sutter T, Killeen T, Gruber P, Petersen JA, Weller M, Linnebank M. Monitoring long-term efficacy of fampridine in gait-impaired patients with multiple sclerosis. Neurology. 2017 Feb 28;88(9):832-841. doi: 10.1212/WNL.0000000000003656. Epub 2017 Feb 1. PMID 28148629
- [Derived] Zorner B, Filli L, Reuter K, Kapitza S, Lorincz L, Sutter T, Weller D, Farkas M, Easthope CS, Czaplinski A, Weller M, Linnebank M. Prolonged-release fampridine in multiple sclerosis: Improved ambulation effected by changes in walking pattern. Mult Scler. 2016 Oct;22(11):1463-1475. doi: 10.1177/1352458515622695. Epub 2016 Jan 13. PMID 26762672